CLINICAL TRIAL: NCT01760044
Title: Noninvasive Assessment of Tissue Perfusion Status in Critically Ill Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kevin Kuo, Fellow, Pediatric Critical Care, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NATP001
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Sepsis; Shock
Keywords: tissue oxygenation; perfusion status
MeSH Terms: conditions — Sepsis; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tissue oxygenation monitoring (Experimental): Tissue oxygenation monitoring
  Interventions: Device: Tissue oxygenation monitoring

INTERVENTIONS:
Device: Tissue oxygenation monitoring — The device provides continuous measures with updates based on the previous 10 seconds worth of data. Data is continuously stored.
  Other Names: R-StO2 (Raman Tissue Oxygenation)

SUMMARY:
Investigators are conducting research about oxygen levels in the body and whether it is possible to use a device to measure oxygen in the body's tissues noninvasively, without blood draws or a catheter (a plastic tube placed in a vein). Investigators would like to know how this device compares to standard measurements using blood from a catheter. This may help treat patients who may not be getting enough oxygen to their body.

DETAILED DESCRIPTION:
Investigators will enroll patients in the pediatric intensive care unit who have an indwelling catheter that allows measurement of central venous oxygen saturation. Measurements of central venous oxygen saturation using blood oximetry will be compared with measures of tissue oxygenation at the buccal mucosa using a Raman spectroscopy tissue oximeter. Investigators will also measure the status of the sublingual microcirculation utilizing sidestream dark field microscopy. Basic demographic and clinical variables such as ongoing vasoactive infusions, mechanical ventilation, and laboratory data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Pediatric Intensive Care Unit (PICU) or Pediatric Cardiothoracic Unit (PCTU)
* Age >30 days and <18 years -patients with a "high" central venous line (ie internal jugular, subclavian, peripherally inserted central catheter, broviac, port) capable of blood draw and with central venous catheter tip in the superior vena cava

Exclusion Criteria:

* Age <30 days or >18 years
* Known pregnancy or subsequently discovered pregnancy after admission
* Uncorrected cyanotic congenital heart disease

Relative Exclusion Criteria:

* Oral trauma preventing placement of Raman StO2 oximeter probe or microcirculation video device
* Upper extremity trauma preventing placement of BEAM device

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation level as measured by raman spectroscopy device | The measures will occur twice within the first 24 hours of admission to the pediatric ICU and then whenever a central venous oxygen saturation is measured by the clinical care team until the patient is discharged from the pediatric ICU.
  Measurement of tissue oxygenation level as based upon raman spectroscopy device will be compared with standard measures from central venous oxygen saturation from central venous catheters.

SECONDARY OUTCOMES:
Microcirculation as recorded by sublingual video microcirculation recorder. | Twice in the first 24 hours after PICU admission
  Two video clips will be recorded of the sublingual microcirculation in each patient within the first 24 hours of admission to the PICU.
Vital signs as recorded by Bioinformatically enabled armband monitor (BEAM) | Continuous from PICU admission through 24 hours of admission
  Bioinformatically enabled armband monitor (BEAM) will be placed on the patient's upper extremity for the first 24 hours of their admission and will be subsequently removed. The data will be stored in the device and investigators and clinicians caring for subjects will be blinded to the device output as data is collected. The device continually captures physiologic data such as heart rate, ECG results, and temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ward, MD, Principal Investigator — University of Michigan
Locations (1):
- C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States